CLINICAL TRIAL: NCT01881737
Title: An Open-Label Pilot Study of Pregnenolone in the Treatment of Individuals With Autism
Brief Title: A Study of Pregnenolone in the Treatment of Individuals With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-08092011-8246
Record Dates: First submitted 2011-11-28; First posted 2013-06-20 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Autistic Disorder
Keywords: autism
MeSH Terms: conditions — Autistic Disorder | interventions — Pregnenolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pregnenolone (Experimental): Pregnenolone up to 500 mg per day
  Interventions: Drug: Pregnenolone

INTERVENTIONS:
Drug: Pregnenolone — With Baseline serving as approximately day 1, twice daily intake of orally administered pregnenolone will occur on a schedule consisting of an up-titration followed by a down-titration as described below.
  Week 1 and 2: 100 mg
  Week 3 and 4: 200 mg
  Week 5 and 6: 300 mg
  Week 7 and 8: 400 mg
  Week 9 -12: 500 mg
  At the end of Week 12, pregnenolone was decreased by 50 mg twice a day every 3 days until it was discontinued.
  If the participant is unable to tolerate a specific dose then he/she will be maintained at the highest tolerated dose until down titration occurs.

SUMMARY:
This study will assess the tolerability and effectiveness of pregnenolone in the treatment of behavioral deficits in adults with autism. Pregnenolone is a naturally occurring hormone found in the body which has been shown to help with the function of nerve cells. It is also shown to modulate the activity of certain brain receptors implicated in autism. We hope to examine the tolerability of pregnenolone in adults with autism.

DETAILED DESCRIPTION:
This study will assess the tolerability and effectiveness of pregnenolone in the treatment of behavioral deficits in adults with autism. Pregnenolone is a naturally occurring hormone found in the body which has been shown to help with the function of nerve cells. It is also shown to modulate the activity of certain brain receptors implicated in autism.

Pregnenolone has been used safely in research studies involving individuals with schizophrenia. In the proposed trial, we hope to examine the tolerability of pregnenolone in adults with autism. We hope to see improvement in behavioral outcomes as measured by standardized behavioral measures. Further, we will measure concentrations of pregnenolone and related neuroactive compounds in the blood. The use of pregnenolone has been studied in a number of mental disorders but not autism. Thus, we hope the study will identify new avenues of research for the treatment of autism.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients 18-45 years of age;
2. Males and females who are physically healthy;
3. Diagnosis of autism based on Diagnostic and Statistical Manual (DSM-IV-TR) criteria, the Autism Diagnostic Interview-Revised, and expert clinical evaluation;
4. Total Aberrant Behavior Checklist (ABC) greater then 21;
5. Care provider who can reliably bring subject to clinic visits, can provide trustworthy ratings, and interacts with subject on a regular basis;
6. Ability of subject to swallow the compound;
7. Stable concomitant medications for at least 2 weeks; and
8. No planned changes in psychosocial interventions during the open-label pregnenolone trial.

Exclusion Criteria:

1. Diagnostic and Statistical Manual (DSM-IV-TR) diagnosis of schizophrenia, schizoaffective disorder, or psychotic disorder, not otherwise specified;
2. Prior adequate trial of pregnenolone;
3. Active medical problems: unstable seizures, significant physical illness (e.g., serious liver or renal pathology);
4. Pregnancy or sexually active females (as determined by a urinary pregnancy test in the beginning of the study); and
5. Subjects taking oil or fat based nutritional supplements will be excluded from the study unless they have been off these compounds for at least 4 weeks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Fung LK, Libove RA, Phillips J, Haddad F, Hardan AY. Brief report: an open-label study of the neurosteroid pregnenolone in adults with autism spectrum disorder. J Autism Dev Disord. 2014 Nov;44(11):2971-7. doi: 10.1007/s10803-014-2144-4. PMID 24849255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between November 2011 and September 2013 at Stanford University.
Groups:
- Pregnenolone: Open-Label Trial
Period: Overall Study
Arm/Group | Pregnenolone
Started | 15 (This is a pilot study)
Number Screened | 15
Completed | 10
Not Completed | 5
Not completed — Inclusion/Exclusion Criteria Not Met | 3
Not completed — Withdrawal by Subject | 1
Not completed — Worsening of baseline behavior | 1

BASELINE CHARACTERISTICS:
Population: 15 subjects were consented; however, 3 of those subjects did not meet the inclusion/exclusion requirements so they could not participate in the trial and were not included in the baseline analysis population.
Groups:
- Pregnenolone: Twice daily intake of orally administered pregnenolone will occur on a schedule consisting of an up-titration followed by a down-titration as described below.
  Week 1 and 2: 100 mg Week 3 and 4: 200 mg Week 5 and 6: 300 mg Week 7 and 8: 400 mg Week 9 -12: 500 mg At the end of Week 12, pregnenolone was decreased by 50 mg twice a day every 3 days until it was discontinued.
  If the participant is unable to tolerate a specific dose then he/she will be maintained at the highest tolerated dose until down titration occurs.
Arm/Group | Pregnenolone
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events According to Dosage Record and Treatment Emergent Symptom (DOTES) as Assessed at All Follow-up Visits (2, 4, 6, 8, 10, 12, and 16 Weeks)
Time Frame: 2, 4, 6, 8, 10, 12, and 16 weeks
Population: During the 12-week treatment period, two participants dropped out of the study. The follow-up observations for the two participants who dropped out were included in the analyses.
Measure: Number; unit: participants
Groups:
- Pregnenolone: Open-Label study
Arm/Group | Pregnenolone
Number analyzed (Participants) | 12
participants
  Tiredness | 1
  Diarrhea | 2
  Depressive Affect | 2
  Increased Excitement/Agitation | 3
  Sleep Problems | 1
  Drowsiness | 1
  Anorexia/Decreased Appetite | 2
  Increased Motor Activity | 1
  Sweating | 1
  Constipation | 1
  Tremor | 1

2. Secondary Outcome: Social Responsiveness Scale (SRS) Total Score
Description: SRS total score (total range 0-195); higher scores mean more abnormal social behaviors.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: SRS total score (total range 0-195)
Groups:
- Pregnenolone: Pregnenolone up to 500 mg per day
  Pregnenolone: With Baseline serving as approximately day 1, twice daily intake of orally administered pregnenolone will occur on a schedule consisting of an up-titration followed by a down-titration as described below.
  Week 1 and 2: 100 mg
  Week 3 and 4: 200 mg
  Week 5 and 6: 300 mg
  Week 7 and 8: 400 mg
  Week 9 -12: 500 mg
  At the end of Week 12, pregnenolone was decreased by 50 mg twice a day every 3 days until it was discontinued.
  If the participant is unable to tolerate a specific dose then he/she will be maintained at the highest tolerated dose until down titration occurs.
Arm/Group | Pregnenolone
Number analyzed (Participants) | 12
SRS total score (total range 0-195)
  Baseline SRS Total Score | 84.9 (8.1)
  Week 12 SRS Total Score | 84.5 (9.2)
Statistical Analysis 1: Comparison: Pregnenolone; Effect Size Cohen's d = -0.05; Test type: Superiority or Other; p = 0.848, Paired t test

3. Secondary Outcome: Sensory Profile Questionnaire Total Score
Description: scores on a scale (range: 38-190); lower scores mean more abnormal sensory problems.
Time Frame: 12
Population: During the 12-week treatment period, two participants dropped out of the study. The follow-up observations for one of the participants who dropped out were included in the analyses.
Measure: Mean (Standard Deviation); unit: scores on a scale (range: 38-190)
Arm/Group | Pregnenolone
Number analyzed (Participants) | 11
scores on a scale (range: 38-190)
  Baseline Score on the Sensory Profile | 137.7 (21.5)
  Week 12 Score on the Sensory Profile | 147.6 (15.3)
Statistical Analysis 1: Comparison: Pregnenolone; Test type: Superiority or Other; p = 0.009, Paired t test; Effect Size Cohen's d = 0.53

4. Secondary Outcome: Vineland Adaptive Behavior Scale
Description: Adaptive Behavior Composite Score (score range 20-160); higher scores mean more typical adaptive behaviors.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score (range 20-160)
Arm/Group | Pregnenolone
Number analyzed (Participants) | 12
score (range 20-160)
  Baseline Vineland Adaptive Behavior Score | 37.3 (13.1)
  Week 12 Vineland Adaptive Behavior Score | 42.9 (16.5)
Statistical Analysis 1: Comparison: Pregnenolone; Test type: Superiority or Other; p = 0.38, paired t test; Effect size Cohen's d = 0.38

5. Secondary Outcome: Repetitive Behavior Scale
Time Frame: 12 weeks
Population: Data were not collected for this Outcome Measure because the total score is not a very valid measure of receptive behaviors.
Arm/Group | Pregnenolone
Number analyzed (Participants) | 0

6. Secondary Outcome: Pregnenolone Level in Peripheral Blood as Measured at Baseline and After 12 Weeks
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Pregnenolone
Number analyzed (Participants) | 11
ng/ml
  Baseline level | 1.9 (0.7)
  Week 12 | 7.0 (4.1)
Statistical Analysis 1: Comparison: Pregnenolone; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Time Frame: Baseline, 2, 4, 6, 8, 10, 12, and 16 weeks
Groups:
- Pregnenolone: Pregnenolone was not associated with any severe adverse effects. Single episodes of tiredness (n = 1), diarrhea (n = 1), and depressive affect (n = 1) that could possibly be related to pregnenolone were reported. A few other adverse events with remote chance to be related to the medication were reported: increased excitement/agitation (n = 3), sleep problems (n = 1), drowsiness (n = 1), anorexia/decreased appetite (n = 2), increased motor activity (n = 1), sweating (n = 1), constipation (n = 1), diarrhea (n = 1), tremor (n = 1), and depressive affect (n = 1). No significant vital sign or EKG changes occurred in any study participants. No abnormal laboratory tests were caused by pregnenolone.
Arm/Group | Pregnenolone
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnenolone (N=12)
Tiredness (General disorders) | 1 (1) — Single episode of tiredness (n = 1) that could possibly be related to pregnenolone was reported.
Diarrhea (Gastrointestinal disorders) | 2 (2) — Single episode of diarrhea (n = 1) that could possibly be related to pregnenolone and a single episode (n = 1) with remote chance to be related were reported.
Depressive Affect (Psychiatric disorders) | 2 (2) — Single episodes of depressive affect (n = 1) that could possibly be related to pregnenolone and a single episode (n = 1) with a remote chance to be related were reported.
Increased Excitement/Agitation (Psychiatric disorders) | 3 (3) — Single episodes of excitement/agitation (n = 3) with a remote chance to be related to the medication were reported.
Sleep Problems (General disorders) | 1 (1) — Single episode of sleep problems (n = 1) with remote chance to be related to the medication was reported.
Drowsiness (General disorders) | 1 (1) — Single episode of drowsiness (n = 1) with a remote chance to be related to the medication was reported.
Anorexia/Decreased Appetite (Gastrointestinal disorders) | 2 (2) — Single episodes of anorexia/decreased appetite (n = 2) with a remote chance to be related to the medication were reported.
Increased Motor Activity (General disorders) | 1 (1) — Single episode of increased motor activity (n = 1) with a remote chance to be related to the medication was reported.
Sweating (General disorders) | 1 (1) — Single episode of sweating (n = 1) with a remote chance to be related to the medication was reported.
Constipation (Gastrointestinal disorders) | 1 (1) — Single episode of constipation (n = 1) with a remote chance to be related to the medication was reported.
Tremor (General disorders) | 1 (1) — Single episode of tremor (n = 1) with a remote chance to be related to the medication was reported.

LIMITATIONS AND CAVEATS:
This is an open-label trial with a very small sample size. No measures of plasma or salivary concentrations of metabolites were completed in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No